CLINICAL TRIAL: NCT06980220
Title: Impact of Perineal Massage With Lubricating Gel During Expulsion on Perineal Outcomes
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier de Gonesse (Other)
Responsible Party: Sponsor
Other Study IDs: 0043_MATERNITE
Record Dates: First submitted 2025-05-12; First posted 2025-05-20 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Perineal Massage; Perineum/Injuries; Labor, Obstetric; Episiotomy
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The primary goal is to assess whether this practice reduces the incidence and severity of perineal tears. Secondary objectives include evaluating the impact of the massage on perineal pain in the postpartum period and on the episiotomy rate. Participants will include primiparous women with singleton pregnancies who delivered spontaneously via vaginal birth. Exclusion criteria include instrumental deliveries, breech presentations, and preterm births. Data will be collected through a questionnaire filled out by midwives immediately after birth, as well as additional data extracted from medical records. All data will be anonymized using a birth number code. The questionnaire collects information on whether a perineal massage was performed, the type of product used, the birth position, use of warm compresses, performance of the Ritgen maneuver, and perineal outcomes. The medical record will provide demographic and clinical data, including the mother's age, BMI, labor duration, pushing time, newborn weight, and head circumference. The study aims to provide evidence on whether perineal massage with gel at expulsion is an effective strategy to prevent severe perineal trauma and improve postpartum recovery.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy
* Spontaneous vaginal delivery
* Primiparous women (first-time mothers)

Exclusion Criteria:

* Instrumental births
* In-seat births
* Premature births

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: The study will select participants from primiparous women (first-time mothers) who have delivered through spontaneous vaginal births at the hospital. The population will consist of women with singleton pregnancies who are undergoing vaginal delivery without any complications requiring instrumental intervention or preterm delivery. The study will focus on a cohort of women who have received care from midwives, ensuring consistency in the delivery approach. Participants will be selected based on the inclusion criteria outlined and will be monitored for perineal outcomes, including the occurrence of perineal tears and postpartum pain.
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2023-10-15 (Actual); Primary Completion 2024-05-15 (Actual); Study Completion 2024-05-15 (Actual)

PRIMARY OUTCOMES:
Rate of Perineal Tears Following Perineal Massage with Lubricating Gel at Expulsion | 15/10/2023 - 15/05/2024

CONTACTS AND LOCATIONS:
Locations (1):
- France, Gonesse, France